CLINICAL TRIAL: NCT04021979
Title: Comparison of Two Bowel Cleansing Regimens（Controlled Dietary Restriction With Enteral Nutrition and 1.5L Polyethylene Glycol vs Controlled Dietary Restriction and 2.0L Polyethylene Glycol）：an Endoscopist-blinded, Prospective Randomized Controlled Trial
Brief Title: Effectiveness of Enteral Nutrition for Dose Reduction of Low Dose PEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2017-R035
Record Dates: First submitted 2019-07-05; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Bowel Preparation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral Nutritional+PEG (Experimental): Enteral Nutritional Powder with low volume 1.5L PEG
  Interventions: Dietary Supplement: Enteral Nutrition Powder Ensure; Drug: 1.5L PEG
- Self-controlled diet+PEG (Placebo Comparator): Self-controlled diet with normal amount of 2L PEG
  Interventions: Other: Self-controlled diet; Drug: 2L PEG

INTERVENTIONS:
Dietary Supplement: Enteral Nutrition Powder Ensure — Enteral Nutrition Powder Ensure for each meal.The duration of study is one day before colonoscopy.
  Other Names: Ensure
  Arms: Enteral Nutritional+PEG
Drug: 1.5L PEG — Low volume PEG
  Other Names: Hengkangzhengqing
  Arms: Enteral Nutritional+PEG
Other: Self-controlled diet — Self-controlled low residue diet.
  Arms: Self-controlled diet+PEG
Drug: 2L PEG — Normal volume of PEG
  Other Names: Hengkangzhengqing
  Arms: Self-controlled diet+PEG

SUMMARY:
This clinical trial is being conducted to assess whether dietary restriction with enteral nutrition prescribed could prevent nonadherence to dietary restrictions, enable additional reduction of the required volume of PEG-ELS.

DETAILED DESCRIPTION:
Bowel preparation plays a vital role in the quality of colonoscopy.Bowel preparation consists of 2 key steps: dietary restriction and purgative ingestion.Two liters of PEG-ELS are widely used in Asian countries, but in a well-designed clinical trial，additional reduction of PEG-ELS volume seems feasible. Enteral nutrition may simplify the process and avoid unexpected intake of fiber-containing food.

We hypothesized that dietary restriction with enteral nutrition prescribed could prevent nonadherence to dietary restrictions, enable additional reduction of the required volume of PEG-ELS.

ELIGIBILITY:
Inclusion Criteria:

1. the age of 18-75year
2. Outpatients undergoing colonoscopy
3. Informed consent

Exclusion Criteria:

1. the age >75 years or <18 years
2. history of colectomy or bowel obstruction
3. severe constipation (defined as stool frequerncy of 3 or less/week)
4. current pregnancy or breastfeeding
5. BMI >30, diabetes
6. known allergies to cleansing agents or ingredients of Enteral nutrition
7. inability to follow the oral bowel preparation regimen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
the quality of bowel preparation | 1day
  Evaluation of the quality of bowel preparation for each participant by the Ottawa bowel preparation scale(OBPS)，it's a validated scoring system with scores between 0 and 14, where 0 is the best score，The score comprises a sub score 0-4 for each colon segment: right, transverse and rectosigmoid colon.n addition, a score 0-2 is added to indicate the total amount of luminal fluid.

SECONDARY OUTCOMES:
patients' satisfaction with the process of bowel preparation | 1day
  At the end of the procedure, the patients were asked about the satisfaction with the process of bowel preparation. Satisfaction includes bad，not so bad and good.Bad means that the patient is not satisfied with the program, not so bad means that the patient is satisfied with the plan, and good means that the patient is very satisfied with the plan.
patients' willingness to have the colonoscopy done again at this facility in the future | 1day
  It represent participants who wanted to choose the same protocol in the future as they received in this trial.Including yes and no two options, if yes, indicating that the patient is willing to undergo colonoscopy again, if no, indicating that the patient is reluctant to undergo colonoscopy again.
comparison with previous experience | 1day
  If patients with colonoscopy times ≥ 2, they need to compare with previous experience，Including better than last experience, similar to the last experience, and worse than the last experience.
adverse events | 1day
  It represent the incidence of abdominal cramping, bloating, nausea/vomiting after intake of PEG and/or enteral nutrition was compared.
Convenience of Protocol between enteral nutrition with low volume 1.5L PEG and Self-controlled diet with normal amount of 2L PEG Protocol | 1day
  It represented the percentage of patients who thinks the protocol is easy to use.

CONTACTS AND LOCATIONS:
Overall Officials: Hongpeng Lu, master, Principal Investigator — Department of Gastroenterology, Ningbo No. 1 Hospital, Ningbo, China
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No